CLINICAL TRIAL: NCT03773900
Title: Characterization of Gut Microbiota Composition and Activity After a Daily Supplementation of 4.5 g/Day of ChitinGlucan Fibre During 3 Weeks in At-cardiometabolic Risk Volunteers
Acronym: FITACHITIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 69HCL18_0362
Record Dates: First submitted 2018-11-16; First posted 2018-12-12 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Cardiometabolic Risk; Abdominal Obesity
Keywords: chitin-glucan; gut microbiota; Fecal Short Chain Fatty Acid (SCFA); cardiometabolic risk; nutritional challenge test; biomarkers
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chitin-Glucan supplementation (Experimental)
  Interventions: Dietary Supplement: Kiotransine (chitin-glucan from aspergillus niger)
- Placebo supplementation (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Kiotransine (chitin-glucan from aspergillus niger) — The volunteers will take three times a day one bag of powder containing 1.5g of chitin-glucan fiber during three weeks. The powder will be diluted in water.
  Arms: Chitin-Glucan supplementation
Dietary Supplement: Placebo — The volunteers will take three times a day one bag of powder containing placebo during three weeks. The powder will be diluted in water.
  Arms: Placebo supplementation

SUMMARY:
The aim of this study is to demonstrate the beneficial effects on gut microbiota composition and activity of the diary intake of insoluble fiber (extract from Aspergillus Niger) for three weeks. The first studies about the fiber have shown a favorable gut microbiota modulation and an improvement of metabolic parameters like LDL cholesterol. In addition to fecal measurements, several biomarkers of colic fermentation will be assessed: expired gases, PolyUnsaturated Fatty Acid, Short Chain Fatty Acid (SCFA) after a rich-fiber breakfast (= 15 grams) and a nutritional challenge test at lunch. The gastrointestinal tolerance of fiber intake and the intestinal transit modification will be also followed during all the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-smokers
* Body mass index between 25 and 35 kg/m2
* Waist circumference < 80cm for women and > 94 cm for men
* Fiber intake <25g/day

Exclusion Criteria:

* Medical history of digestive surgery or disease
* Current or recent (<12 weeks) intake of antibiotics or gastro-intestinal medicinal product
* Current probiotics, prebiotics, fiber complement, and/or any products modulation gut transit
* Feeding particular diet such as vegetarian diet or hyperprotein diet
* Current weight loss diet
* Pregnant or lactating woman or woman who did not use effective contraception
* Drinking more than 3 glasses of alcohol per day (>30g/day)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Fecal SCFA | baseline and three weeks
  Change from baseline fecal SCFA at three weeks by Gas chromatography-Flame Ionization Detector

SECONDARY OUTCOMES:
gut microbiota composition | baseline and three weeks
  Change from baseline gut microbiota composition by 16SrDNA Illimina Sequencing
fecal biliary acids | baseline and three weeks
  Change from baseline fecal biliary acids by FAME quantification (gas-liquid chromatography)
fecal PolyUnsaturated Fatty Acids (PUFA) | baseline and three weeks
  Change from baseline fecal PolyUnsaturted Fatty Acids (PUFA) by FAME quantification (gas-liquid chromatography)
fecal albumin | baseline and three weeks
  Change from baseline fecal albumin by immunoenzymatic technique (ELISA)
fecal zonulin | baseline and three weeks
  Change from baseline fecal zonulin by immunoenzymatic technique (IDK Zonulin ELISA)
fecal calprotectin | baseline and three weeks
  Change from baseline fecal calprotectin by Phadia 100 system
TLR-agonist in stool | baseline and three weeks
  Change from baseline TRL-agonist in stool using the HEK-Blue™ TLR cellules
Change from baseline CO2, CH4 and H2 kinetics in exhaled gases | baseline and three weeks
  by gas chromatography, during ten hours after rich-fiber breakfast and nutritional challenge test at lunch
body composition | baseline and three weeks
  Change from baseline bodycompositio by bioimpedancemetry
Change from plasma glucose kinetics | baseline and three weeks
  by spectrophotometry method , during seven hours after rich-fiber breakfast and nutritional challenge test at lunch
Change from plasma insulin kinetics | baseline and three weeks
  by radio-immuno analysis , during seven hours after rich-fiber breakfast and nutritional challenge test at lunch
Change from plasma Non-Esterifies Fatty-Acid (NEFA) kinetics | baseline and three weeks
  by spectrophotometry method , during seven hours after rich-fiber breakfast and nutritional challenge test at lunch
plasma TriacylGlycerol (TG) kinetics | baseline and three weeks
  Change from plasma TriacylGlycerol (TG) kinetics by spectrophotometry method , during seven hours after rich-fiber breakfast and nutritional challenge test at lunch
Cholesterol Total, Cholesterol LDL | baseline and three weeks
  Change from baseline cholesterol Total, Cholesterol LDL by spectrophotometry method
resting energy expenditure | baseline and three weeks
  Change from baseline resting energy expenditure by indirect calorimetry
stool consistency | every week, up to three weeks
  by Bristol Stool Chart (type1-7)
stool frequency | every week, up to three weeks
  by questionnaire
gastro-intestinal symptoms | every week, up to three weeks
  by questionnaires and visual analogue scale (VAS) score (on a 90mm horizontal line; from no symptom (minimal) to serious symptom (maximum))
quality of life during the study | baseline and three weeks
  change from baseline quality of life during the study by SF 36 questionnaire
change from baseline dietary intake of fibre | baseline and three weeks
  by three day food record

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche en Nutrition Humaine Rhône-Alpes - Centre hospitalier Lyon Sud, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ranaivo H, Zhang Z, Alligier M, Van Den Berghe L, Sothier M, Lambert-Porcheron S, Feugier N, Cuerq C, Machon C, Neyrinck AM, Seethaler B, Rodriguez J, Roumain M, Muccioli GG, Maquet V, Laville M, Bischoff SC, Walter J, Delzenne NM, Nazare JA. Chitin-glucan supplementation improved postprandial metabolism and altered gut microbiota in subjects at cardiometabolic risk in a randomized trial. Sci Rep. 2022 May 25;12(1):8830. doi: 10.1038/s41598-022-12920-z. PMID 35614185
- See also: Related Info — http://www.crnh-rhone-alpes.fr